CLINICAL TRIAL: NCT00767767
Title: The Effect of Intravenous Anesthetics on Fear Learning and Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0710009434; K08GM083213 (NIH)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Phobias
Keywords: anesthetic drugs, associative memory, fear
MeSH Terms: conditions — Phobic Disorders | interventions — Propofol; Thiopental

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebos (Placebo Comparator): Saline Infusion
  Interventions: Drug: Placebos
- Propofol 0.45mcg/mL (Active Comparator): Anesthetic Drug Infusion
  Interventions: Drug: Propofol 0.45mcg/mL
- Propofol 0.90mcg/mL (Active Comparator): Anesthetic Drug Infusion
  Interventions: Drug: Propofol 0.90mcg/mL
- Thiopental 1.5mcg/mL (Active Comparator): Anesthetic Drug Infusion
  Interventions: Drug: Thiopental 1.5mcg/mL
- Thiopental 3mcg/mL (Active Comparator): Anesthetic Drug Infusion
  Interventions: Drug: Thiopental 3mcg/mL

INTERVENTIONS:
Drug: Placebos — IV Saline infusion for 2 hours.
  Arms: Placebos
Drug: Propofol 0.45mcg/mL — IV Propofol infusion for 2 hours.
  Other Names: Propofol
  Arms: Propofol 0.45mcg/mL
Drug: Propofol 0.90mcg/mL — IV Propofol infusion for 2 hours.
  Other Names: Propofol
  Arms: Propofol 0.90mcg/mL
Drug: Thiopental 1.5mcg/mL — IV Thiopental 1.5mcg/mL infusion for 2 hours
  Other Names: Thiopental
  Arms: Thiopental 1.5mcg/mL
Drug: Thiopental 3mcg/mL — IV Thiopental 3mcg/mL infusion for 2 hours
  Other Names: Thiopental
  Arms: Thiopental 3mcg/mL

SUMMARY:
People often develop fearful responses to things, but have no conscious control over the fear. This is a basic form of unconscious memory, called "fear conditioning." Intravenous anesthetic drugs have remarkable effects on conscious memory, but it is unknown whether they have similar effects on these unconscious fear memories.

To address this question, the investigators will study 114 healthy adult volunteer subjects. The subject is given a very low dose of an anesthetic drug intravenously (i.e. through the bloodstream). The dose is so low that the subject might not even be able tell if they are getting the drug. While they are receiving the drug, the subject will perform a series of memory tests and a fear conditioning experiment, which are set up like a very simple computer game. To create the "fear response", subjects will occasionally receive a mildly uncomfortable shock to their arm. The subject is able to determine the highest level of shock that they will receive.

The investigators are doing this study because the investigators wish to know exactly how the drugs affect the way people process fear and emotion. This knowledge might one day be used in the treatment of some psychiatric disorders.

DETAILED DESCRIPTION:
People often develop fearful responses to things, but have no conscious control over the fear (e.g. phobias). This is a basic form of unconscious memory, called "fear conditioning." Intravenous anesthetic drugs have remarkable effects on conscious memory, but it is unknown whether they have similar effects on these unconscious fear memories.

To address this question, the investigators will study 114 healthy adult volunteer subjects. The subject is given a very low dose of an anesthetic drug intravenously (i.e. through the bloodstream). The dose is so low that the subject might not even be able tell if they are getting the drug. While they are receiving the drug, the subject will perform a series of memory tests and a fear conditioning experiment, which are set up like a very simple computer game. To create the "fear response", subjects will occasionally receive a mildly uncomfortable shock to their arm. The subject is able to determine the highest level of shock that they will receive.

The investigators are doing this study because the investigators wish to know exactly how the drugs affect the way people process fear and emotion. This knowledge might one day be used in the treatment of some psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50
* minimum of high school education
* fluent in English
* normal vocabulary

Exclusion Criteria:

* any significant medical or psychiatric comorbidity (e.g. asthma, diabetes, hypertension, depression, high anxiety)--subjects must be in excellent health such that they would be classified as American Society of Anesthesiologists Physical Status Class I
* deficit in vision or hearing that would impede the study
* allergies to any of the study drugs, to soybeans, or to eggs
* a history of head trauma
* a family history of major psychiatric illness
* body mass index > 30 kg/m2
* a recent history of recreational drug use
* prior exposure to the study materials
* pregnancy
* a personal or family history of any porphyria
* failure to exhibit a skin conductance response to deep inspiration
* the ability to read Chinese characters
* assessment by the investigators that the subject may be unable to cooperate or comply with the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kane Pryor, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol 0.9mcg/mL: Anesthetic Drug Infusion
  Propofol 0.9mcg/mL: IV Propofol infusion for 2 hours.
- Thiopental 1.5mcg/mL: Anesthetic Drug Infusion
  Thiopental 1.5mcg/mL: IV Thiopental infusion for 2 hours.
- Thiopental 3mcg/mL: Anesthetic Drug Infusion
  Thiopental 3mcg/mL: IV Thiopental Infusion for 2 hours.
Period: Overall Study
Arm/Group | Placebos | Propofol 0.45mcg/mL | Propofol 0.9mcg/mL | Thiopental 1.5mcg/mL | Thiopental 3mcg/mL
Started | 21 | 20 | 20 | 3 | 3
Completed | 21 | 20 | 20 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol 0.9mcg/mL: Anesthetic Drug Infusion
  Propofol 0.9mcg/mL: IV Propfol infusion for 2 hours.
- Total: Total of all reporting groups
Arm/Group | Placebos | Propofol 0.45mcg/mL | Propofol 0.9mcg/mL | Thiopental 1.5mcg/mL | Thiopental 3mcg/mL | Total
Number analyzed (Participants) | 21 | 20 | 20 | 3 | 3 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (4.4) | 25.4 (4.1) | 25.6 (4.5) | 23.7 (3.4) | 26.3 (5.8) | 25.2 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 16 | 2 | 0 | 42
  Male | 7 | 10 | 4 | 1 | 3 | 25

OUTCOME MEASURES:

1. Primary Outcome: GSR Trial 1
Description: Galvanic skin repose (GSR) to the first habituation trial (yes/no). Coding: Yes (0) and No (1)
Time Frame: First Trial, for up to 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebos | Propofol 0.45mcg/mL | Propofol 0.9mcg/mL | Thiopental 1.5mcg/mL | Thiopental 3mcg/mL
Number analyzed (Participants) | 21 | 20 | 20 | 3 | 3
units on a scale | .62 (.50) | .55 (.51) | .55 (.51) | .67 (.5) | 0 (0)

ADVERSE EVENTS:
Arm/Group | Placebos | Propofol 0.45mcg/mL | Propofol 0.90mcg/mL | Thiopental 1.5mcg/mL | Thiopental 3mcg/mL
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/20 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/21 | 1/20 | 0/20 | 0/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebos (N=21) | Propofol 0.45mcg/mL (N=20) | Propofol 0.90mcg/mL (N=20) | Thiopental 1.5mcg/mL (N=3) | Thiopental 3mcg/mL (N=3)
Extreme Fidgety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Extremely fidgety, dosing on and off, requiring prompting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes